CLINICAL TRIAL: NCT03823937
Title: Evaluation of Smell and Taste in Patients With Fibromyalgia
Brief Title: Evaluation of Smell and Taste in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: Tugba Ozsoy2
Record Dates: First submitted 2019-01-27; First posted 2019-01-31 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; smell; taste
MeSH Terms: conditions — Fibromyalgia; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: Diagnosed with ACR 2016 criteria
  Interventions: Other: Sniffin' Sticks test and Taste strips
- Control: 18-70 years healthy subjects
  Interventions: Other: Sniffin' Sticks test and Taste strips

INTERVENTIONS:
Other: Sniffin' Sticks test and Taste strips — Sniffin' Sticks test (Burghardt®, Wedel, Germany) is a psychophysical test. It allows semi-objective assessment of the patient's olfactory performance by means of 3 subtests: threshold test, identification test and discrimination test. The Sniffin' Sticks Olfactory Test Kits contain pen like bodies as, for example, in pens used to write on flipcharts or whiteboards.These pen-like bodies, however, contain a fibre stick which is filled with scents. For testing, the cap should be removed so the patient can smell on the tip of the pen.
  The taste strips are a validated examination procedure to investigate the taste ability. When testing the whole mouth taste ability, the taste strips are applied by putting them on the tongue and closing the mouth.

SUMMARY:
Patients diagnosed with fibromyalgia syndrome according to 2016 ACR criteria and 18-70 years old healthy subjects will be included in the study. Their smell and taste will be assessed with sniffin sticks and taste strips. Besides they will be evaluated for quality of life, anxiety, depression, and alexithymia.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of fibromyalgia patients
* Giving informed consent
* Knowing how to write and read in Turkish

Exclusion Criteria:

* Mentally retarded patients
* Psychiatric disorders (bipolar disorder, schizophrenia etc.)
* Severe organ failure (kidney, liver, heart failure)
* History of head trauma
* Any disorder associated with smell and taste functions

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18-70 years old fibromyalgia diagnosed with 2016 ACR criteria and age, sex-matched healthy controls will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hur K, Choi JS, Zheng M, Shen J, Wrobel B. Association of alterations in smell and taste with depression in older adults. Laryngoscope Investig Otolaryngol. 2018 Feb 21;3(2):94-99. doi: 10.1002/lio2.142. eCollection 2018 Apr. PMID 29721540
- [Background] Lotsch J, Kraetsch HG, Wendler J, Hummel T. Self-ratings of higher olfactory acuity contrast with reduced olfactory test results of fibromyalgia patients. Int J Psychophysiol. 2012 Nov;86(2):182-6. doi: 10.1016/j.ijpsycho.2012.09.003. Epub 2012 Sep 15. PMID 22985737

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibromyalgia: Diagnosed with ACR 2016 criteria
  Sniffin' Sticks test and Taste strips: Sniffin' Sticks test (Burghardt®, Wedel, Germany) is a psychophysical test. It allows semi-objective assessment of the patient's olfactory performance by means of 3 subtests: threshold test, identification test and discrimination test. The Sniffin' Sticks Olfactory Test Kits contain pen like bodies as, for example, in pens used to write on flipcharts or whiteboards.These pen-like bodies, however, contain a fibre stick which is filled with scents. For testing, the cap should be removed so the patient can smell on the tip of the pen.
  The taste strips are a validated examination procedure to investigate the taste ability. When testing the whole mouth taste ability, the taste strips are applied by putting them on the tongue and closing the mouth.
- Control: 18-70 years healthy subjects
  Sniffin' Sticks test and Taste strips: Sniffin' Sticks test (Burghardt®, Wedel, Germany) is a psychophysical test. It allows semi-objective assessment of the patient's olfactory performance by means of 3 subtests: threshold test, identification test and discrimination test. The Sniffin' Sticks Olfactory Test Kits contain pen like bodies as, for example, in pens used to write on flipcharts or whiteboards.These pen-like bodies, however, contain a fibre stick which is filled with scents. For testing, the cap should be removed so the patient can smell on the tip of the pen.
  The taste strips are a validated examination procedure to investigate the taste ability. When testing the whole mouth taste ability, the taste strips are applied by putting them on the tongue and closing the mouth.
Period: Overall Study
Arm/Group | Fibromyalgia | Control
Started | 30 | 20
Completed | 30 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia | Control | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (8.47) | 45.65 (9.95) | 45.86 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.07 (5.37) | 26.04 (4.24) | 27.26 (5.01)

OUTCOME MEASURES:

1. Primary Outcome: Sniffin' Sticks Test Score
Description: total smell test score minimum score: 0 maximum score: 48 Higher scores reflect better smell function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia | Control
Number analyzed (Participants) | 30 | 20
score on a scale | 25.96 (6.50) | 36.40 (4.50)

2. Primary Outcome: Taste Strips Test Score
Description: total taste score minimum score: 0 maximum score: 16 Higher scores indicate better taste function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia | Control
Number analyzed (Participants) | 30 | 20
score on a scale | 9.93 (2.65) | 13.55 (1.76)

3. Secondary Outcome: Quality of Life Score
Description: A EQ-5D-3L is a standardized instrument for measuring generic health status. minimum score: -0.59 maximum score: 1 Higher scores indicate better health status.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia | Control
Number analyzed (Participants) | 30 | 20
score on a scale | 0.452 (0.288) | 0.916 (0.109)

4. Secondary Outcome: Anxiety Score
Description: Hamilton anxiety scale: Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia | Control
Number analyzed (Participants) | 30 | 20
score on a scale | 21.23 (9.22) | 5.45 (4.24)

5. Secondary Outcome: Alexithymia Score
Description: Toronto alexithymia scale minimum score: 20 maximum score: 100 Cut-off scores: ≤50=no alexithymia, 51-60=borderline alexithymia, and ≥61=alexithymia
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia | Control
Number analyzed (Participants) | 30 | 20
score on a scale | 57.20 (13.12) | 46.80 (11.30)

6. Secondary Outcome: Depression Score
Description: Hamilton depression scale is designed to rate the severity of depression in patients. Although it contains 21 areas, calculate the patient's score on the first 17 answers.
  Minimum score:0 Maximum score: 53 Higher scores reflect more severe depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia | Control
Number analyzed (Participants) | 30 | 20
score on a scale | 18.03 (7.75) | 5.70 (5.98)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed
Arm/Group | Fibromyalgia | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03823937/Prot_SAP_000.pdf